CLINICAL TRIAL: NCT04569071
Title: A Multi-center Clinical Trial to Evaluate the Efficacy and Safety of MRI-guided Laser Interstitial Thermal Therapy for Medical Refractory Epilepsy
Brief Title: Clinical Trial of MgLiTT for Medical Refractory Epilepsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); Peking Union Medical College Hospital (Other); Chinese PLA General Hospital (Other); Peking University International Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HK593202002
Record Dates: First submitted 2020-09-10; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Epilepsy
Keywords: Stereotactic surgery; Thermal ablation; Medical refractory epilepsy; Epilepsy surgery
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sinovation Laser Ablation System treatment (Experimental): Sinovation Laser Ablation System treatment
  Interventions: Device: Sinovation Laser Ablation System

INTERVENTIONS:
Device: Sinovation Laser Ablation System — In the present single arm study. All eligible subjects will undergo MgLiTT with the Sinovation Laser Ablation System.

SUMMARY:
Multicenter, open-label, prospective designed study to characterize the performance of MRI-guided laser interstitial thermal therapy (MgLiTT) using the Sinovation Laser Ablation System for the treatment of medical refractory epilepsy.

DETAILED DESCRIPTION:
The Sinovation Laser Ablation System uses robot-assisted, precise, high-intensity laser light to initiate necrosis of abnormal brain tissue through thermal ablation while limiting injury to adjacent healthy tissue. MgLiTT has the advantages of precision, minimal invasive procedure and real-time thermal monitoring.

Subjects who meet the study eligibility criteria and sign the informed consent form will undergo the MgLiTT procedure. Subjects, or their caregivers, are required to keep a seizure diary throughout the study, beginning after surgery. The study will monitor and record subjects' seizure frequency, antiepileptic medications, and physical and emotional health.

Subjects treated with Sinovation Laser Ablation System will have at least 9 months of follow-up. Throughout study participation, the study investigator will continuously monitor and document both effectiveness and safety data at study appointments.

ELIGIBILITY:
Inclusion Criteria:

* The age ranged from 6 months to 70 years old;
* Previous diagnosis of drug-resistant epilepsy with focal lesions;
* The average seizure frequency was more than 2 times/month within 3 months;
* Surgical treatment is suitable for epilepsy;
* The subjects or their guardians can understand the purpose of the trial, show adequate compliance with the trial protocol, and sign the informed consent form.

Exclusion Criteria:

* MRI contraindication;
* Patients with severe coagulation dysfunction;
* Pregnant or lactating women;
* Subjects who have participated in clinical trials of any other drugs or medical devices within 3 months;
* Evidence of severe or uncontrollable systemic diseases, as judged by the researchers;
* Subjects considered unsuitable for the clinical trial.

Ages: 6 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-08-08 (Actual); Primary Completion 2021-05-08 (Estimated); Study Completion 2022-02-08 (Estimated)

PRIMARY OUTCOMES:
MgLiTT ablation rate | Within 3 days after operation
  Measurement of postsurgical MRI

SECONDARY OUTCOMES:
Seizure free rate | 90±7 days after operation
  Follow-up
Seizure reduction rate | 90±7 days after operation
  Follow up
Operation time | Within 1 day after operation
  Medical recording
Postsurgical hospitalization | Within 1 day after discharged from hospital
  Medical recording
Mini-Mental State Examination (MMSE) score | Before and 90±7 days after operation
  Range from 0 to 30; Lower score indicates worse cognitive impairment
Quality of life in epilepsy-31 inventory (QOLIE-31) score | Before and 90±7 days after operation
  For adult; Range from 0 to 100; Higher score indicates better quality of life
Quality of life in epilepsy for Adolescents (QOLIE-AD-48) score | Before and 90±7 days after operation
  For Adolescents; Range from 0 to 100; Higher score indicates better quality of life
Vital signs-body temperature | Before and 2±1 days after operation
  From medical recording; Centigrade
Vital signs-pulse | Before and 2±1 days after operation
  From medical recording; Times/minute
Vital signs-respiratory rate | Before and 2±1 days after operation
  From medical recording; Times/minute
Vital signs-blood pressure | Before and 2±1 days after operation
  From medical recording; Systolic pressure/diastolic pressure (mmHg)

OTHER OUTCOMES:
Instrument performance evaluation | Within 1 day after operation
  Higher score indicates better instrument performance
The amount of bleeding | During operation
  Medical recording
Postsurgical complication rates | Within 1 day after discharged from hospital
  Medical recording
Failure free rate of laser ablation minimally invasive treatment kit | Within 1 day after operation
  Medical recording
Failure rate of magnetic resonance guided laser ablation system | Within 1 day after operation
  Medical recording
Incidence of adverse events and serious adverse events | Within 1 day after discharged from hospital
  Medical recording

CONTACTS AND LOCATIONS:
Overall Officials: Kai Zhang, Dr., Study Director — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
We may only share clinical information (rather privacy information) in academic or other reasonable request.
Supporting Information: Analytic Code
Time Frame: After the clinical trials.
Access Criteria: reasonable requests.